CLINICAL TRIAL: NCT06259045
Title: Cardiac Cachexia in Advanced Heart Failure - a Prospective Cohort Study Investigating Prevalence and Outcome
Brief Title: Cardiac Cachexia in Advanced Heart Failure
Acronym: CACH-IT-AHF
Status: Active, not recruiting | Type: Observational
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 334613
Record Dates: First submitted 2024-01-26; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Advanced Heart Failure; Cardiac Cachexia; Weight Loss
Keywords: Advanced heart failure; Cardiac cachexia; Heart failure; Unintentional weight loss; Frailty; Sarcopaenia; Cachexia
MeSH Terms: conditions — Weight Loss; Heart Failure; Frailty; Cachexia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Advanced heart failure: Patients enrolled will all have advanced heart failure, defined by a set criteria

SUMMARY:
Heart failure is a condition in which the heart stops pumping effectively, causing symptoms such as breathlessness or leg swelling. It affects around 900,000 people in the United Kingdom. As our population gets older, this number will continue rise. It is a condition with poor overall survival - nearly 50% of patients die within 5 years of being diagnosed with heart failure.

Cardiac cachexia is a complex condition associated with heart failure. There is general loss of muscle with or without loss of fat in cardiac cachexia. The main feature of cardiac cachexia is therefore unintentional weight loss in heart failure patients. The reason why it develops is poorly understood currently. Importantly, some studies have shown that cardiac cachexia is more likely to lead to poorer outcomes (such as death) in the patients who develop it.

However, there have been no studies, to our knowledge, that look at this condition in those patients who have very weak hearts ('advanced heart failure').

The investigators are looking to clarify how common cardiac cachexia is within advanced heart failure patients, and secondly how outcomes compare to those advanced heart failure patients that do not have the condition. With this in mind, the investigators will be able to establish the fuller impact cardiac cachexia has on survival and outcomes in patients with advanced heart failure. This study will involve assessing a group of ~200 advanced heart failure patients for cardiac cachexia to establish an estimate of how common it is overall. The investigators will then follow up the patients over a year, to see if we can assess the impact of cardiac cachexia on survival and outcomes.

Overall, the investigators therefore hope this study will give a more robust picture on the true impact of cardiac cachexia in advanced heart failure. By doing so, the investigators will firstly highlight its importance to other clinicians who will better be able to monitor and or diagnose it, and secondly pave way for more research on a potential treatment strategy for this condition.

DETAILED DESCRIPTION:
Cardiac cachexia (CC) is a complex metabolic syndrome associated with chronic heart failure, characterised by loss of muscle with or without loss of fat. The prominent clinical feature of CC is unintentional weight loss in adults. Anorexia, inflammation, insulin resistance and increased muscle protein breakdown are frequently associated with wasting disease. Cachexia is associated with increased morbidity, is infrequently identified or diagnosed and rarely treated. Using an older definition of CC, previous studies have found its presence to confer a poorer overall prognosis (50% mortality at 18 months follow-up in a cohort of general heart failure patients). Depending on the definition used, the prevalence of CC in heart failure has been described in literature as anywhere between 10 - 37%. The pathogenesis of CC is poorly understood, but is likely to be multi factorial, driven by a low cardiac output resulting in an increase in catabolic versus anabolic metabolism.

A consensus definition from 2008 now states that CC is present when a patient has non-oedematous weight loss of at least 5% in ⩽12 months or body mass index <20 kg/m2, plus three out of five other criteria including: (i) Decreased muscle strength (ii) Fatigue (iii) Anorexia (iv) Low fat-free mass index (v) Abnormal biochemistry e.g. Increased inflammatory markers (C-reactive protein, interleukin-6), anaemia, or low serum albumin.

The prevalence of CC in advanced heart failure (AHF), however, has not been described. In this cohort of patients, independent prognosticators are vitally important given the overall propensity towards deterioration and morality. AHF refers to those patients at the end of the clinical spectrum of heart failure. There are a number of criteria to identify patients with AHF, one of which being the 'I NEED HELP' criteria.

The investigators hypothesise that the prevalence of CC in AHF confers a poorer prognosis when compared to the general heart failure population. By establishing its true prevalence and prognostic impact in AHF, the group aim to highlight the need to diagnose cardiac cachexia in AHF earlier, so patients can undergo the appropriate level of closer monitoring and/or escalation in terms of potential invasive therapies or cardiac transplantation where appropriate.

This study will involve participants with AHF being recruited from a single tertiary cardiac centre, via both inpatient and outpatient settings. Participants will be assessed for CC using the aforementioned 2008 CC criteria. After study enrollment, eligible participants will undergo follow up over 12 months'. This will allow the investigators to evaluate the prevalence and 12-month prognosis of cardiac cachexia in an advanced heart failure population in a hospital setting.

ELIGIBILITY:
Inclusion Criteria:

* Meets one of the "I NEED HELP" markers for advanced heart failure
* Has capacity to consent and participate in the study
* Age 18 years and older

Exclusion Criteria:

* Does not have at least one "I NEED HELP" marker for advanced heart failure
* Does not consent to or has not got the ability to participate in the study
* Is below the age of 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced heart failure are being recruited in to this study
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-01-25 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Combined composite primary end point of: all-cause mortality or cardiac transplantation or left ventricular assist device (LVAD) insertion | 12 months
  This combined composite primary end-point will assess for multiple adverse outcomes within our cohort, which will be assessed for and combined to form this single primary end point. If the participants were to: die due to any cause, undergo cardiac transplantation or LVAD insertion over the 12 month follow-up period, then the primary end-point will have been reached. Comparisons will be made between participants with and without cardiac cachexia in our cohort.

SECONDARY OUTCOMES:
Hospitalisation secondary to heart failure | 12 months
  If participants were hospitalised secondary to heart failure causes over the 12 month follow up period, they will have reached this end-point. Comparisons will be made between patients with and without cardiac cachexia in our cohort.
New ventricular arrhythmogenesis | 12 months
  If participants develop any ventricular arrhythmia over the 12 month follow up period, they will have reached this end-point. Comparisons will be made between participants with and without cardiac cachexia in our cohort.
New stroke | 12 months
  If participants develop a stroke within the 12 month follow up period, they will have reached this end-point. Comparisons will be made between participants with and without cardiac cachexia in our cohort.
New myocardial Infarction | 12 months
  If participants develop a myocardial infarction within the 12 month follow up period, they will have reached this end-point. Comparisons will be made between participants with and without cardiac cachexia in our cohort.
Cardiovascular death | 12 months
  If participants die secondary to a cardiovascular cause within the 12 month follow up period, they will have reached this end-point. Comparisons will be made between participants with and without cardiac cachexia in our cohort.
Hospitalisation (all-cause) | 12 months
  If participants were hospitalised for any reason over the 12 month follow up period, they will have reached this end-point. Comparisons will be made between patients with and without cardiac cachexia in our cohort.
Changes to quality of lifestyle questionnaire KCCQ-12 | 12 months
  Changes to the Kansas city cardiomyopathy Questionnaire-12 (KCCQ-12) score from baseline to 12 months will be assessed. Comparisons will be made between patients with and without cardiac cachexia in our cohort.
Changes to quality of lifestyle questionnaire MLWHFQ | 12 months
  Changes to the Minnesota Living with Heart Failure Questionnaire (MLWHFQ) score from baseline to 12 months will be assessed. Comparisons will be made between patients with and without cardiac cachexia in our cohort.

CONTACTS AND LOCATIONS:
Locations (1):
- Harefield Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
TBC